CLINICAL TRIAL: NCT02303860
Title: Pharmacokinetic Study of ORM-12741 After Multiple Oral Doses
Brief Title: Pharmacokinetic Study of Multiple Doses of ORM-12741 (Nebula PK 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3098013
Record Dates: First submitted 2014-10-21; First posted 2014-12-01 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Healthy volunteer study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Panel 1 (Experimental): Adaptive design: Each subject will receive MR A or MR B formulation of ORM-12741 or a combination of these once or twice daily for one week either combined with IR formulation or not.
  Interventions: Drug: ORM-12741 MR A; Drug: ORM-12741 MR B; Drug: ORM-12741 IR
- Panel 2 (Experimental): Adaptive design: Each subject will receive MR A or MR B formulation of ORM-12741 or a combination of these once or twice daily for one week either combined with IR formulation or not.
  Interventions: Drug: ORM-12741 MR A; Drug: ORM-12741 MR B; Drug: ORM-12741 IR

INTERVENTIONS:
Drug: ORM-12741 MR A — Modified release formulation of ORM-12741
Drug: ORM-12741 MR B — Modified release formulation of ORM-12741
Drug: ORM-12741 IR — Immediately release formulation of ORM-12741

SUMMARY:
The purpose of this study is to evaluate ORM-12741 concentrations in blood at steady state.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate pharmacokinetic and safety of ORM-12741 after multiple oral dosing of modified release formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Good general health ascertained by detailed medical history and physical examination.
3. Females and males between 18 and 65 years of age (inclusive).
4. Body mass index (BMI) between 18-30 kg/m2 (inclusive, BMI = weight/height2).
5. Weight 50-100 kg (inclusive).
6. Regular intestinal transit (no recent history of recurrent constipation, diarrhoea, or other intestinal problems).

Exclusion Criteria:

1. Predicted poor compliance or inability to communicate well with the investigator or the study centre personnel.
2. Veins unsuitable for repeated venipuncture or cannulation.
3. Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
4. Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. Hormonal contraception and hormone replacement therapy are allowed.
5. Susceptibility to severe allergic reactions.
6. Intake of any medication that could affect the outcome of the study, within 2 weeks prior to the first study treatment administration or less than 5 times the half-life of the medication. Possible enzyme inducing drugs will be discussed case-by-case with the sponsor.
7. Regular consumption of more than 21 units of alcohol per week for males and 16 units per week for females (1 unit = 4 cl spirits, about 13 g of alcohol).
8. Current use of nicotine-containing products more than 5 cigarettes or equivalent/day.
9. Inability to refrain from using nicotine-containing products during the stay at the study centre.
10. Inability to refrain from consuming caffeine-containing beverages during the stay at the study centre, e.g. propensity to develop headaches when refraining from caffeine-containing beverages.
11. Blood donation or loss of significant amount of blood within 3 months prior to the first study treatment administration.
12. Any clinically significant 12-lead electrocardiogram (ECG) abnormality after 10-minute rest in supine position at the screening visit, as judged by the investigator. For example:

    - QTc (calculated with the Bazett's formula) > 470 msec for females and 450 msec for men.
13. HR < 45 beats/minute or > 100 beats/minute after a 10-minute rest in supine position at the screening visit.
14. At the screening visit systolic blood pressure (BP) < 90 mmHg or > 150 mmHg after a 10- minute rest in supine position, diastolic BP < 50 mmHg or > 90 mmHg after a 10-minute rest in supine position, or symptomatic orthostatic hypotension, or

    * decrease of ≥ 20 mmHg of systolic BP or
    * decrease of ≥ 10 mmHg of diastolic BP after 3 minutes in standing position.
15. Any abnormal value in laboratory tests, or vital signs, or physical examination finding, which in the opinion of the investigator could interfere with the interpretation of the test results or cause a health risk for the subject if he takes part in the study.
16. History of drug abuse or positive result in drug abuse test.
17. Positive serology to human immunodeficiency virus antibodies (HIVAgAb), hepatitis C virus antibodies (HCVAb) or hepatitis B surface antigen (HBsAg).
18. Females of childbearing potential if they are not using proper contraception (hormonal contraception, intrauterine device [IUD] or surgical sterilization, spermicidal foam in conjunction with condom on male partner) during the study. Use of oral/hormonal contraception alone is not acceptable. (Note: women of childbearing potential with no current heterosexual relationship can be included without contraception according to the judgement of the investigator).
19. Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk for the study subject.
20. Participation in a clinical drug study within 3 months prior to the first study treatment administration of this study or earlier participation in a clinical study with ORM-12741.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, AUC, T1/2 | Blood samples collected once at day 2, 4, 6, 9, 10 and 11; twice on day 8 and frequently on day 7.
  Pharmacokinetics

SECONDARY OUTCOMES:
Safety - adverse events, vital signs, ECG, safety laboratory values | 8 days per treatment period
  Adverse events, vital signs, ECG, safety labs

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, Principal Investigator — Clinical Research Services Turku - CRST Oy
Locations (1):
- Clinical Research Services Turku - CRST Oy, Turku, Finland